CLINICAL TRIAL: NCT02244489
Title: A Phase 1b Study Evaluating Momelotinib Combined With Capecitabine and Oxaliplatin in Subjects With Relapsed/Refractory Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Momelotinib Combined With Capecitabine and Oxaliplatin in Adults With Relapsed/Refractory Metastatic Pancreatic Ductal Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-370-1369
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Relapsed/Refractory Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Recurrence | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Momelotinib (MMB)+capecitabine (Experimental): Participants will receive momelotinib (MMB)+capecitabine at varying dose levels to determine the MTD for momelotinib (MMB) and capecitabine.
  Interventions: Drug: Momelotinib (MMB); Drug: Capecitabine
- Momelotinib (MMB)+capecitabine+oxaliplatin (Experimental): Upon reaching the MTD for momelotinib (MMB) and capecitabine or if no MTD is reached, participants will receive momelotinib (MMB)+capecitabine at the MTD plus oxaliplatin at varying dose levels to determine the MTD of combination capecitabine, momelotinib (MMB), and oxaliplatin.
  Interventions: Drug: Momelotinib (MMB); Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Momelotinib (MMB) — Momelotinib (MMB) tablet(s) administered orally once or twice daily
  Other Names: GS-0387; CYT387
Drug: Capecitabine — Capecitabine tablet(s) administered orally twice daily for 14 days, followed by 7 days off, until the end of treatment
Drug: Oxaliplatin — Oxaliplatin administered intravenously over 120 minutes or as per institutional standard of care on Day 1 of each 21-day cycle.
  Arms: Momelotinib (MMB)+capecitabine+oxaliplatin

SUMMARY:
This study will evaluate the safety, tolerability, and define the maximum tolerated dose (MTD) of momelotinib (MMB) combined with capecitabine and oxaliplatin in adults with relapsed/refractory metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

* Relapsed or refractory metastatic pancreatic adenocarcinoma
* Received 1 prior chemotherapy regimen for metastatic pancreatic ductal adenocarcinoma (not including neoadjuvant and/or adjuvant therapy)
* Measurable disease per RECIST v1.1
* Adequate organ function defined as

  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x upper limit of normal (ULN) OR ≤ 5 x ULN if liver metastases are present; total conjugated bilirubin ≤ 2 x ULN
  * Absolute neutrophil count (ANC) ≥1500 cells/mm^3, platelet ≥100,000 cells/mm^3, hemoglobin ≥ 9.0 g/dL
  * Creatinine clearance (CrCl) > 50 ml/min as calculated by the Cockroft-Gault method
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Key Exclusion Criteria:

* Received more than 1 prior line of chemotherapy for metastatic pancreatic ductal adenocarcinoma
* Major surgery within 21 days of first dose of study drug
* Minor surgical procedure(s) within 7 days of enrollment or not yet recovered from prior minor surgery (placement of central venous access device, fine needle aspiration, or endoscopic biliary stent ≥ 1 day before enrollment is acceptable)
* Chemotherapy, immunotherapy, biologics, and/or investigational therapy within 21 days prior to first dose of study drug
* Known positive status for HIV, chronic active or acute viral hepatitis A, B, or C infection, or hepatitis B or C carrier
* Known dihydropyrimidine dehydrogenase deficiency
* Peripheral neuropathy ≥ Grade 2
* Any condition that impairs gastrointestinal absorption of drug
* Known or suspected brain or central nervous system metastases
* Diagnosis of pancreatic islet neoplasm, acinar cell carcinoma, non-adenocarcinoma, adenocarcinoma originating from the biliary tree or cystadenocarcinoma
* External biliary drain
* Documented myocardial infarction or unstable/uncontrolled cardiac disease within 6 months of enrollment

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | Up to 21 days
  Dose limiting toxicities refer to toxicities experienced during the first 21 days of treatment that have been judged to be clinically significant and at least possibly related to study treatment.
Incidence of adverse events, assessment of clinical laboratory test findings, physical examination, 12-lead electrocardiogram (ECG), and vital signs measurements | Up to 2 years
  This composite endpoint will measure the safety profile of momelotinib.

SECONDARY OUTCOMES:
Overall response rate | Up to 2 years
  Overall response rate (ORR) is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) as assessed by the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Overall survival | Up to 2 years
  Overall survival (OS) is defined as the interval from first dose date of study drug to death from any cause.
Progression-free survival | Up to 2 years
  Progression-free survival (PFS) is defined as the interval from first dose date of study drug to the earlier of the first documentation of definitive disease progression or death from any cause; definitive disease progression is progression based on RECIST criteria v1.1.
Pharmacokinetic (PK) profile of momelotinib (MMB) | Predose and postdose on Day 15
  This composite endpoint will measure the plasma PK profile of momelotinib (MMB). The following parameters will be measured, where applicable:
  * Cmax: maximum observed concentration of drug in plasma
  * Ctau: observed drug concentration at the end of the dosing interval
  * AUCtau: concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (4):
- United States (4):
  - Scottsdale Healthcare Research Institute, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Tennessee Oncology, Nashville, Tennessee
  - Virginia Cancer Specialists, PC, Fairfax, Virginia